CLINICAL TRIAL: NCT07238634
Title: Comparative Effects of Dynamic Movement Intervention and Bobath Approach on Neuromuscular Development in Spastic Cerebral Palsy
Brief Title: Effects of DMI vs Bobath on Neuromuscular Development in CP
Acronym: DMINDTSCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Prof. Dr. Shoaib Waqas, Professor, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBS24LMSPT027
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Dynamic Movement Intervention; Bobath Therapy
Keywords: Dynamic Movement Intervention; Bobath Therapy; Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Interventional Study Model: Randomized Clinical Trial (Parallel-Group Design):
  This study will adopt a randomized clinical trial (RCT) model, employing a parallel-group design to evaluate and compare the effects of two physiotherapeutic interventions-Dynamic Movement Intervention (DMI) and the Bobath (Neurodevelopmental) Approach-on neuromuscular development in children with spastic cerebral palsy.
  Participants who meet the inclusion criteria will be randomly assigned into two groups:
  Group A (Experimental Group): will receive Dynamic Movement Intervention (DMI). Group B (Control Group): will receive therapy based on the Bobath Approach. Both groups will undergo intervention sessions of equal duration and frequency under standardized conditions. Pre- and post-intervention assessments will be conducted using validated neuromuscular and functional outcome measures to ensure objectivity.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Dynamic Movement Intervention
- Group B (Active Comparator)
  Interventions: Other: Bobath Therapy

INTERVENTIONS:
Other: Dynamic Movement Intervention — Participants will receive Dynamic Movement Intervention (DMI) consisting of task-specific, structured, repetitive, and progressively challenging exercises designed to improve neuromuscular control. The intervention will be delivered for 12 weeks, with evaluations at baseline (week 0), mid-intervention (week 6), and post-intervention (week 12). DMI sessions will include dynamic tasks such as rolling on soft or unstable surfaces to promote trunk rotation and segmental control; sitting balance training on therapy balls or foam pads with perturbations to activate trunk and head righting responses; and trunk stability exercises in quadruped and kneeling positions to enhance coordination and proprioception. Standing activities on balance discs or BOSU balls will target weight shifting, small squats, and multidirectional reaching for balance control, while walking tasks on varied surfaces(foam mats, tactile paths and beams)will challenge gait, coordination, and postural alignment.
  Arms: Group A
Other: Bobath Therapy — Participants in this group will receive therapy based on the Bobath Concept (Neurodevelopmental Treatment), an evidence-informed, problem-solving approach designed to facilitate normal movement patterns, inhibit abnormal tone, and improve postural control and functional mobility in children with spastic cerebral palsy. The intervention will be implemented over 12 weeks, with evaluations at baseline (week 0), mid-intervention (week 6), and post-intervention (week 12). The Bobath approach emphasizes individualized handling and facilitation techniques aimed at enhancing postural alignment, balance reactions, and coordinated functional movements. The therapist uses guided facilitation at key points of control-such as the pelvis, trunk, and shoulders-to promote normal movement synergies and reduce the influence of spasticity or abnormal reflex patterns.
  Arms: Group B

SUMMARY:
Cerebral palsy (CP) is a leading cause of permanent motor disability in children, resulting from non-progressive disturbances to the developing brain. Prematurity and low birth weight are major risk factors, with infants under 1500 g having a markedly higher risk. Spastic CP is the most common subtype, and spastic diplegia accounts for 30-40% of cases, primarily affecting the lower limbs and trunk control. CP prevalence has declined in high-income countries but remains higher in low- and middle-income regions, including Pakistan. Beyond clinical challenges, CP imposes a substantial lifelong economic burden. Current management follows the ICF framework, emphasizing function, participation, and independence. Traditional approaches such as the Bobath method show limited evidence compared with task-oriented therapies. Dynamic Movement Intervention (DMI) is a neuroplasticity-based, task-oriented approach emphasizing repetitive functional activities. Trunk-focused dynamic training has shown superior improvements in balance and gross motor function. However, comparative evidence between DMI and Bobath therapy in young children is limited, necessitating further research using validated outcome measures.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a major cause of permanent motor disability in childhood and is defined as a group of non-progressive disorders affecting movement and posture due to disturbances in the developing fetal or infant brain. Its etiology is multifactorial, with prematurity and low birth weight identified as the strongest risk factors. Population-based European studies indicate that infants weighing less than 1500 g at birth have up to a 70-fold greater risk of developing CP compared with those born weighing over 2500 g.

Spastic CP is the most prevalent subtype, with spastic diplegia accounting for approximately 30-40% of cases. This subtype primarily affects the lower extremities and is characterized by increased muscle tone, poor trunk control, and persistent limitations in functional mobility. Clinical presentation varies from isolated motor deficits in focal brain injury to complex impairments involving sensory, cognitive, communicative, and behavioral domains when brain involvement is extensive.

Recent meta-analyses report a decline in CP prevalence in high-income countries to approximately 1.6 per 1,000 live births, whereas substantially higher rates, up to 3.4 per 1,000 live births, persist in low- and middle-income countries. In Pakistan, regional data from Khyber Pakhtunkhwa report a prevalence of 1.22 per 1,000 live births, with a male predominance. Beyond clinical impact, CP imposes a considerable economic burden, with estimated lifetime costs exceeding USD 860,000 per affected individual.

Current CP management aligns with the International Classification of Functioning, Disability, and Health (ICF) framework, emphasizing activity, participation, and functional independence. Although early intervention benefits cognitive outcomes, sustained improvements in motor function remain inconsistent. Traditional neurodevelopmental approaches, particularly the Bobath method, focus on tone regulation and movement facilitation; however, systematic reviews indicate limited evidence supporting their superiority over task-oriented therapies. Consequently, contemporary guidelines advocate for evidence-based, goal-directed interventions that yield meaningful functional outcomes.

Dynamic Movement Intervention (DMI) is a task-based therapeutic approach grounded in neuroplasticity principles, emphasizing repetitive, progressive, and functionally relevant activities. Given the proximal-to-distal pattern of motor development, trunk control is fundamental for balance, coordination, and mobility. Evidence suggests that trunk-focused training on dynamic surfaces enhances postural control, sensory integration, and gross motor function more effectively than static surface exercises. Task-oriented training further promotes motor learning through repetition of meaningful activities, facilitating adaptive reorganization of motor pathways.

Randomized trials and systematic reviews support the effectiveness of trunk-targeted and task-oriented interventions in improving trunk stability, balance, and gross motor function in children with CP. However, direct comparisons between DMI and the Bobath approach remain limited, particularly in young children with spastic diplegic CP. Moreover, the Trunk Impairment Scale (TIS), a validated predictor of functional mobility, has been underutilized as a primary outcome measure. This study aims to address these gaps by comparing the effects of DMI and Bobath therapy on neuromuscular development in children aged 2-4 years with spastic diplegic CP using validated outcome measures, including the GMFM-88, SSDT, and TIS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spastic diplegic cerebral palsy.
* Gross Motor Function Measurement Scale (GMFC) level I to III.
* Children who have head control.
* Ability to understand and follow simple instructions.

Exclusion Criteria:

* Visual or hearing impairments (e.g., cataract, myopia, deafness).
* Cognitive problems impacting participation.
* Uncontrolled convulsions or recent seizure activity.
* Orthopedic surgeries of the lower limbs, such as dorsal rhizotomy within the last year.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure-88 (GMFM-88) | 12 weeks
  A standardized observational tool used to assess changes in gross motor function across five dimensions, including lying, sitting, crawling, standing, and walking, specifically designed for children with cerebral palsy.
Shoaib Sensorimotor Development Tool (SSDT) | 12 weeks
  A specialized tool designed to assess sensorimotor development in children, including sensory integration, motor planning, and coordination. It provides insight into neuromotor function beyond gross motor skills.
Trunk Impairment Scale (TIS) | 12 weeks
  Evaluates trunk control through assessments of static sitting balance, dynamic sitting balance, and trunk coordination. It is essential for measuring core stability and postural control improvements.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghurki Trust Teaching Hospital, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Result] Park EY, Kim WH. Effect of neurodevelopmental treatment-based physical therapy on the change of muscle strength, spasticity, and gross motor function in children with spastic cerebral palsy. J Phys Ther Sci. 2017 Jun;29(6):966-969. doi: 10.1589/jpts.29.966. Epub 2017 Jun 7. PMID 28626301
- [Result] Sah AK, Balaji GK, Agrahara S. Effects of Task-oriented Activities Based on Neurodevelopmental Therapy Principles on Trunk Control, Balance, and Gross Motor Function in Children with Spastic Diplegic Cerebral Palsy: A Single-blinded Randomized Clinical Trial. J Pediatr Neurosci. 2019 Jul-Sep;14(3):120-126. doi: 10.4103/jpn.JPN_35_19. Epub 2019 Sep 27. PMID 31649770